CLINICAL TRIAL: NCT05706948
Title: Effects of High Intensity Interval Training on Cardiopulmonary Parameters With or Without Facemask in Healthy Participants
Brief Title: High Intensity Interval Training on Cardiopulmonary Parameters With or Without Facemask in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC/01370 Muneeba Fatima Tariq
Record Dates: First submitted 2023-01-22; First posted 2023-01-31 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Healthy
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training (With Face Mask) (Experimental)
  Interventions: Other: High Intensity Interval Training (With Face Mask)
- High Intensity Interval Training (Without Face Mask) (Experimental)
  Interventions: Other: High Intensity Interval Training (Without Face Mask)

INTERVENTIONS:
Other: High Intensity Interval Training (With Face Mask) — High Intensity Interval Training on Treadmill for 4 weeks with Face mask
  Arms: High Intensity Interval Training (With Face Mask)
Other: High Intensity Interval Training (Without Face Mask) — High Intensity Interval Training on Treadmill for 4 weeks with out Face mask
  Arms: High Intensity Interval Training (Without Face Mask)

SUMMARY:
To determine the effects of high intensity interval training on cardiovascular function, cardio metabolic markers and cardiorespiratory fitness in healthy individuals with or without facemask

ELIGIBILITY:
Inclusion Criteria:

* Non smoker
* Free of any heart and lung diseases
* Passed Physical Activity Readiness Questionnaire PAR-Q
* To be able to do exercise

Exclusion Criteria:

* Any physical limitation that restrict exercise
* Any neurological illness

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Pulse | 4 weeks
  Changes from the baseline, Pulse will be measured in Beats per minutes with Pulse oximeter.
Oxygen saturation | 4 weeks
  Changes from the baseline, Oxygen saturation will be measured in Percentages with pulse oximeter
Waist circumference | 4 weeks
  Waist circumference will be measured for abdominal or central fat mass. It is measured in cm at the middle distance between the last floating rib and the iliac crest using a retractable ergonomic measuring tape. Change from the baseline to 4 week will be compared
Modified BORG Scale | 4 weeks
  The Modified Borg Dyspnea Scale is numerical rating scale ranging from 0 to 10 and is used to measure dyspnea that patient report during sub-maximal exercise and is regularly administered during six-minute walk test. Changes from the baseline will be measured
Vo2 Max | 4 weeks
  Changes from the baseline ;The maximum or optimum rate at which the heart, lungs and muscles can effectively use oxygen during exercise, used as a way of measuring a person's individual aerobic capacity.
Body Mas Index | 4 weeks
  Changes from the baseline, Body Mass Index can be define as statistical index utilizing an individual's height and weight to give an estimation of muscle versus fat in female and male of all ages. It is determined by taking an individual weight in kilograms, separated by their height in meters squared, or BMI = weight (in kg)/height (in m square).
Hip circumference | 4 weeks
  Hip measurement is an estimation of the hips, utilizing a measuring tape, for assessment of spatial distance between each relating hipbone with respect to the buttocks. Hip circumference can be a significant estimation in deciding combined muscle to fat ratio around the waist that might reflect sedentary lifestyle.
Waist to hip ratio | 4 weeks
  Waist to hip ratio is defined as a ratio of circumference of waist to that of hip.
Forced Expiratory Volume in 1 second (FEV1) | 4 weeks
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 4 weeks
  Changes From the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters.
Peak Expiratory Flow | 4 weeks
  Changes From the Baseline, the digital spirometer is used in clinical setting to analyze Peak Expiratory Flow in Liters.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Islamabad Medical & Surgical Hospital, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No